CLINICAL TRIAL: NCT01294748
Title: Clinical Investigation of a DES (MiStent™ System) With Sirolimus and a Bioabsorbable Polymer for the Treatment of Patients With De Novo Lesions in Native Coronary Arteries.
Brief Title: Clinical Investigation of the MiStent Drug Eluting Stent (DES) in Coronary Artery Disease
Acronym: DESSOLVE-II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Micell Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MIS-CEM-2010-02
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Results first posted 2014-03-26 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2016-12

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Drug-eluting Stent; Sirolimus
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MiStent DES (Experimental): The MiStent SES is a sirolimus-eluting absorbable polymer stent for coronary artery revascularization.
  Interventions: Device: MiStent DES
- Endeavor DES (Active Comparator): The Endeavor DES is an everolimus-eluting durable polymer stent for coronary artery revascularization.
  Interventions: Device: Endeavor DES

INTERVENTIONS:
Device: MiStent DES — The MiStent is a device/drug combination comprised of two components; a stent and a drug product (sirolimus within an absorbable polymer coating).
  Arms: MiStent DES
Device: Endeavor DES — The Endeavor is a device/drug combination comprised of two components; a stent and a drug product (everolimus within a durable polymer coating).
  Arms: Endeavor DES

SUMMARY:
The DESSOLVE II clinical trial is to assess the safety and performance of the sirolimus-eluting MiStent for the treatment for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to discrete de novo lesions in the native coronary arteries.

DETAILED DESCRIPTION:
The DESSOLVE II clinical trial is to assess the safety and performance of the sirolimus-eluting MiStent as compared to the Endeavor DES for the treatment for improving coronary luminal diameter in patients with symptomatic ischemic heart disease due to discrete de novo lesions in the native coronary arteries.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 and ≤85 years;
2. Stable/unstable angina pectoris (Class I-IV), documented ischemia/silent ischemia;
3. Planned single, de novo, types A, B1 or B2 coronary lesions;
4. Target lesion located in a native coronary artery;
5. Target lesion in vessel ranging from 2.5 to 3.5 mm amenable to treatment (coverage) with a 30 mm long stent;
6. Target lesion with >50% diameter stenosis;
7. Recent Q-wave (>72 hours) or non-Q-wave myocardial infarction;
8. Patients eligible for PCI;
9. Candidate for CABG ;
10. A patient may have one additional critical non-target lesion.
11. Patient capable of providing informed consent and is willing to comply with all study requirements.

Exclusion Criteria:

1. Female patients of childbearing potential who do not have a confirmed negative pregnancy test at baseline and are not on some form of birth control;
2. Recent Q-wave MI < 72 hours prior to the index procedure.
3. Recent Q- or non-Q-wave MI with still elevated levels of cardiac markers (e.g. CK; and CK-MB if the CK is elevated);
4. LVEF <30% (within the previous 6-months);
5. Patients in cardiogenic shock;
6. CVA or TIA within the past 6 months;
7. Active GI bleeding within past 3 months;
8. Any prior anaphylactic reaction to contrast agents;
9. Chemotherapy within 30-days before or after the index procedure;
10. Receiving oral or intravenous immunosuppressive therapy or has known life-limiting immunosuppressive or autoimmune disease;
11. Renal dysfunction (creatinine > 2.0 mg/dL or 177 µmol/L);
12. Platelet count <100,000 cells/mm³ or >700,000 cells/mm³;
13. White blood cell count <3,000 cells/mm3;
14. Hepatic disease;
15. Heart transplant recipient;
16. Known contraindication to DAPT;
17. Known hypersensitivity to sirolimus, cobalt-chromium, or to medications such as aspirin, heparin and Angiomax (bivalirudin), and all three of the following: clopidogrel bisulfate (Plavix), ticlopidine (Ticlid), and Prasugrel (Effient);
18. Life expectancy less than 12 months;
19. Any major medical condition that may interfere with participation in this study;
20. Patient is currently participating in an investigational drug or another device study and has not completed the follow-up to the primary endpoint, or the patient is planning on participating prior to completing 12-months follow-up;
21. Target vessel has been treated within 10 mm proximal or distal to target lesion with any type of PCI or within a year prior to index procedure;
22. Planned or actual target vessel(s) treatment with an unapproved device, directional or rotational coronary atherectomy, laser, cutting balloon, or transluminal extraction catheter prior to stent placement;
23. Patient previously treated at any time with brachytherapy;
24. Planned coronary angioplasty or CABG in the first 9 months after the index procedure or any other planned intervention within 30-days post index procedure;
25. Prior PCI of a non-target vessel must be at least 14 days prior to study enrollment;
26. The intent to direct stent the target lesion;
27. Angiographic Exclusion Criteria:

    * In-stent restenotic target lesion;
    * In-stent restenotic target lesion;
    * More than one lesion requiring treatment in the target vessel);
    * Target vessel diameter <2.5 mm or >3.5 mm;
    * Long target lesion not amenable to treatment with up to a 30 mm long stent;
    * Left main critical disease (≥50% DS);
    * Target lesion is located in a surgical bypass graft;
    * Total target vessel occlusion (TIMI flow grade 0-1);
    * Target lesion ostial location;
    * Target lesion at bifurcation involving side branch >2.5 mm or lateral branch that also requires stenting;
    * Calcified target lesion that anticipates unsuccessful/impracticable predilation;
    * Target vessel with excessive tortuosity or proximal angulation;
    * Thrombus present in target vessel;
    * More than one non-target critical lesion;
    * Non-target lesion to be treated during the index procedure meets any of the following criteria:

      1. Located within the target vessel;
      2. Located within a bypass graft ;
      3. Left main location;
      4. Chronic total occlusion
      5. Involves a complex bifurcation.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2011-02; Primary Completion 2012-06 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Wijns, MD, Principal Investigator — Cardiovascular Center, Onze-Lieve-Vrouwziekenhuis Aalst (OLV Hospital)
Locations (28):
- Belgium (6):
  - Cardiovascular Center, Aalst
  - Antwerp Hospital, ZNA Middelheim, Antwerp
  - Brussels University Hospital, Brussels
  - Ziekenhuis Oost-Limburg, Genk
  - Virga Jesse Ziekenhuis, Hasselt
  - KUL Cardiology Gasthuisberg, Leuven
- France (3):
  - Jacques Cartier Hospital, Massy
  - Claude Galien Hospital, Quincy
  - Clinique Pasteur, Toulouse
- Netherlands (5):
  - OLV, Amsterdam
  - St. Antonius Ziekenhuis, Nieuwegein
  - TweeSteden Ziekenhuis, Tilburg
  - UMC Utrecht, Utrecht
  - Hospital Weezenlanden, Zwolle
- New Zealand (5):
  - Auckland City Hospital, Auckland
  - Mercy Angiography Unit, Auckland
  - Christchurch Hospital, Christchurch
  - Dunedin Hospital, Dunedin
  - Wellington Hospital, Wellington
- Sweden (2):
  - Sahlgrenska University Hospital, Gothenburg
  - Orebro University Hospital, Örebro
- United Kingdom (7):
  - Royal Sussex Hosp, Brighton
  - Papworth Hospital, Cambridge
  - Guy's & St. Thomas', London
  - Royal Brompton, London
  - University Hospital South Manchester, Manchester
  - Norfolk/Norwich UHosp, Norwich
  - Southampton UHT, Southampton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rusinaru D, Vrolix M, Verheye S, Chowdhary S, Schoors D, Di Mario C, Desmet W, Donohoe DJ, Ormiston JA, Knape C, Bezerra H, Lansky A, Wijns W; DESSOLVE II Investigators. Bioabsorbable polymer-coated sirolimus-eluting stent implantation preserves coronary vasomotion: A DESSOLVE II trial sub-study. Catheter Cardiovasc Interv. 2015 Dec 1;86(7):1141-50. doi: 10.1002/ccd.25610. Epub 2015 Sep 22. PMID 25044635
- [Derived] Wijns W, Vrolix M, Verheye S, Schoors D, Slagboom T, Gosselink M, Benit E, Donohoe D, Knape C, Attizzani GF, Lansky AJ, Ormiston J; DESSOLVE II Investigators. Randomised study of a bioabsorbable polymer-coated sirolimus-eluting stent: results of the DESSOLVE II trial. EuroIntervention. 2015 Apr;10(12):1383-90. doi: 10.4244/EIJY14M05_03. PMID 24801119

RESULTS

PARTICIPANT FLOW:
Groups:
- Endeavor DES: MiStent DES: The MiStent is a device/drug combination comprised of two components; a stent and a drug product (sirolimus within an absorbable polymer coating).
Period: Overall Study
Arm/Group | MiStent DES | Endeavor DES
Started | 123 | 61
Completed | 118 (At 270 days) | 59 (At 270 days)
Not Completed | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Endeavor DES: Active Comparator: Endeavor DES
- Total: Total of all reporting groups
Arm/Group | MiStent DES | Endeavor DES | Total
Number analyzed (Participants) | 123 | 61 | 184
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.96 (10.43) | 65.13 (10.47) | 65.02 (10.42)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 33 | 94
  >=65 years | 62 | 28 | 90
Gender [Count of Participants; unit: Participants]
  Female | 38 | 16 | 54
  Male | 85 | 45 | 130
Region of Enrollment [Number; unit: participants]
  France | 7 | 3 | 10
  Belgium | 82 | 42 | 124
  Netherlands | 15 | 7 | 22
  United Kingdom | 10 | 5 | 15
  New Zealand | 4 | 3 | 7
  Sweden | 5 | 1 | 6

OUTCOME MEASURES:

1. Primary Outcome: In-Stent Late Lumen Loss
Description: Measured by the angiographic core laboratory as the difference between the post-procedure MLD in the treated segment (stented region) minus the MLD in the same region at follow-up
Time Frame: 9 months
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 103 | 52
mm | 0.27 (0.46) | 0.58 (0.41)

2. Primary Outcome: Major Adverse Cardiac Events (MACE)
Description: Defined as death, MI (Qwave and non-Q-wave) and TVR at 9 months post-procedure. Assessed on all patients with adequate follow-up at 270 days.
Time Frame: 9 months
Measure: Number; unit: percentage of participants
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 117 | 60
percentage of participants | 4.3 [-11.9 to 4.4] | 6.7 [-11.9 to 4.4]

3. Secondary Outcome: Device Success
Description: Achievement of a final in-stent residual diameter stenosis of <50% (by QCA), using the assigned device only.
Time Frame: 8 hours
Measure: Number; unit: percentage of participants
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 122 | 61
percentage of participants | 100 | 100

4. Secondary Outcome: Lesion Success
Description: Achievement of a final in-stent residual diameter stenosis of <50% (by QCA) using any percutaneous method.
Time Frame: 8 hours
Measure: Number; unit: percentage of participants
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 122 | 61
percentage of participants | 100 | 100

5. Secondary Outcome: Procedural Success
Description: Achievement of a final in-stent residual diameter stenosis of <50% (by QCA) using the assigned device (including any adjunctive devices) without cardiac death, MI or repeat revascularization of the target lesion pre-hospital discharge.
Time Frame: 8 hours
Measure: Number; unit: percentage of participants
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 122 | 61
percentage of participants | 98.4 | 96.7

6. Secondary Outcome: Total Mortality
Time Frame: 9-months
Measure: Number; unit: percentage of patients
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 117 | 60
percentage of patients | 0.9 | 1.7

7. Secondary Outcome: Total Myocardial Infarct (MI)
Description: 1. Q-wave MI (QWMI): requires one of the following criteria: development of new abnormal Q waves in ≥2 contiguous ECG leads not present on the patient's baseline (i.e., before intervention) in association with a >2x ULN elevation of CK levels; chest pain or other acute symptoms consistent with myocardial ischemia and new pathological Q waves in ≥2 contiguous ECG leads in the absence of timely cardiac enzyme data.
  2. Non-Q-wave MI (NQWMI):the elevation of CK levels (≥2 times ULN) with elevated CK-MB enzyme levels (≥3 times ULN) in the absence of new pathologic Q waves.
  3. Peri-Procedural MI post PCI:Q or non-Q-wave MI, as defined above, prior to hospital discharge, or CK-MB elevation >3xULN within 48 hours post -PCI, with a normal CK-MB at baseline.
Time Frame: 9-months
Measure: Number; unit: percentage of patients
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 117 | 60
percentage of patients | 2.6 | 3.3

8. Secondary Outcome: Clinically-driven Target Lesion Revascularization (TVR)
Description: TVR is defined as any repeat percutaneous intervention or surgical bypass of any segment of the target vessel (main branch or side branch). The target vessel is defined as the entire major coronary vessel proximal and distal to the target lesion, which includes upstream and downstream branches, and the target lesion itself.
Time Frame: 9-months
Measure: Number; unit: percentage of patients
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 117 | 60
percentage of patients | 0.9 | 3.3

9. Secondary Outcome: Target Vessel Failure (TVF)
Description: Composite endpoint of cardiac death, target-vessel myocardial infarction (Q wave or non-Q wave), and clinically indicated target vessel revascularization
Time Frame: 9-months
Measure: Number; unit: percentage of patients
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 117 | 60
percentage of patients | 3.4 | 6.7

10. Secondary Outcome: Target Lesion Failure (TLF)
Description: Composite endpoint of cardiac death, target-lesion myocardial infarction (Q wave or non-Q wave), and clinically indicated target lesion revascularization
Time Frame: 9-months
Measure: Number; unit: percentage of patients
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 123 | 61
percentage of patients
  TLF to 30 days | 1.7 | 3.3
  TLF to 180 days | 2.5 | 5
  TLF to 270 days | 3.4 | 5

11. Secondary Outcome: Stent Thrombosis (Definite/Probable)
Description: The presence of an intracoronary thrombus that originates in the stent or in the segments 5 mm proximal or distal to the stent post-procedure
Time Frame: 9-months
Measure: Number; unit: percentage of patients
Arm/Group | MiStent DES | Endeavor DES
Number analyzed (Participants) | 117 | 60
percentage of patients | 0 | 1.7

ADVERSE EVENTS:
Time Frame: 270 days
Arm/Group | MiStent DES | Endeavor DES
Serious Adverse Events (participants affected / at risk) | 53/123 | 19/61
Other Adverse Events (participants affected / at risk) | 47/123 | 36/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiStent DES (N=123) | Endeavor DES (N=61)
decompensation cordis (Cardiac disorders) | 1 (1) | 0 (0)
dyspnoe (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
lungoedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
cardiac chest pain (Cardiac disorders) | 1 (1) | 0 (0)
silent ischemia (Cardiac disorders) | 1 (1) | 0 (0)
pneumonia (Infections and infestations) | 1 (1) | 0 (0)
STEMI anterior (caused by acute stent thrombosis) (Cardiac disorders) | 1 (1) | 0 (0)
acute in-stent thrombosis in mid-lad (General disorders) | 1 (1) | 0 (0)
stable angina (Cardiac disorders) | 1 (1) | 2 (2)
angina pectoris (Cardiac disorders) | 1 (1) | 0 (0)
respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
reversible renal failure due to dehydration (Renal and urinary disorders) | 1 (1) | 0 (0)
diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
sudden death (General disorders) | 1 (1) | 0 (0)
accidental fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
inguinal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
in-stent restonosis (Vascular disorders) | 1 (1) | 0 (0)
hip fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
coronary instent restenosis of a non-target lesion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
burning feeling (non-cardiac retrosternal) (General disorders) | 0 (0) | 1 (1)
bleeding at catherer site (General disorders) | 0 (0) | 1 (1)
stenosis left arteria carotis interna (Nervous system disorders) | 1 (1) | 0 (0)
angina (Cardiac disorders) | 1 (1) | 0 (0)
cardiac decompensation (Cardiac disorders) | 0 (0) | 2 (2)
atypical chest pain (Cardiac disorders) | 0 (0) | 1 (1)
occlusions left arteria femoralis (Vascular disorders) | 1 (1) | 0 (0)
femoral pseudo-aneursym (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
coronary silent ischemia (Cardiac disorders) | 1 (1) | 0 (0)
thoracic dyscomfort at exercise (non-cardiac) (General disorders) | 1 (1) | 0 (0)
atypical thoracic pain (General disorders) | 1 (1) | 0 (0)
non-cardiac chest pain (General disorders) | 2 (2) | 3 (3)
angina complaints (Cardiac disorders) | 1 (1) | 0 (0)
subcutaneous bleeding A. Femoralis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ischemic colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
necrotic small bowel (Gastrointestinal disorders) | 0 (0) | 1 (1)
sick sinus syndrome (Cardiac disorders) | 2 (2) | 0 (0)
increasing angina (Cardiac disorders) | 1 (1) | 0 (0)
severe stenosis of distal rca (Cardiac disorders) | 1 (1) | 0 (0)
aorta stenosis just above (Vascular disorders) | 1 (1) | 0 (0)
severe claudication (Vascular disorders) | 1 (1) | 0 (0)
thrombosys of canal of hunter (Vascular disorders) | 1 (1) | 0 (0)
cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
hemorrargic gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
non Q-wave myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
stenosis of arterial iliaca left (Vascular disorders) | 0 (0) | 1 (1)
epigastric bleed due to ulcers (General disorders) | 0 (0) | 1 (1)
restonosis in target vessel, proximal in-stent (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
spiral dissection from mid lad to the most distal (Cardiac disorders) | 0 (0) | 1 (1)
retroperitonial bleeding at femoral bifurcation (Gastrointestinal disorders) | 1 (1) | 0 (0)
RDA prox. stenose (proximally from the stent) (Cardiac disorders) | 1 (1) | 0 (0)
drop in hemoglobin (Investigations) | 1 (1) | 0 (0)
cardiac related chest pain (Cardiac disorders) | 0 (0) | 1 (1)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
psuedoanerysm (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
aortic dissection complicated with anastomosis aorta (Vascular disorders) | 1 (1) | 0 (0)
stenosis de novo (Cardiac disorders) | 0 (0) | 1 (1)
restonosis intrastent 1st diagnoal + proxLAD stenos (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
atrial ventribular block type III (Cardiac disorders) | 1 (1) | 0 (0)
instent restenosis in RCA proximal (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
postprocedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiStent DES (N=123) | Endeavor DES (N=61)
angina pectoris (Cardiac disorders) | 13 (13) | 9 (9)
myocardial infarction (Cardiac disorders) | 0 (0) | 4 (4)
catherer site hematoma (General disorders) | 7 (7) | 5 (5)
chest pain (General disorders) | 0 (0) | 3 (3)
non-cardiac chest pain (General disorders) | 13 (13) | 8 (8)
headache (Nervous system disorders) | 7 (7) | 4 (4)
dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 3 (3)
hypertension (Vascular disorders) | 7 (7) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less